CLINICAL TRIAL: NCT05516719
Title: Longitudinal Investigation of Imidazoline-2 Binding Site as a Novel Marker of Disease Progression in Parkinson's Disease: An [11C]BU99008 PET Study
Brief Title: Longitudinal Investigation of I2BS in PD
Acronym: FOX_2
Status: Recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-21-15
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's; Parkinson Disease; Parkinson's Disease; Neurodegenerative Diseases; Neurodegeneration; Positron Emission Tomography
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Nerve Degeneration | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biosamples collected during this study will be blood, urine, and CSF. Blood biomarkers include routine clinical laboratory, DNA testing, and other analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- SNCA (Alpha-synuclein gene): PET and SPECT molecular imaging and MRI; Clinical investigation and computerized neuropsychological testing; Collection of blood, urine and CSF biomarkers of PD pathology
  Interventions: Other: Positron Emission Tomography (PET) scan using BU99008 tracer; Other: FP-CIT Single-photon Emission Computed Tomography (SPECT) scan; Other: Magnetic Resonance Imaging (MRI) Scan; Other: Lumbar puncture
- Idiopathic Parkinson's Disease: PET and SPECT molecular imaging and MRI; Clinical investigation and computerized neuropsychological testing; Collection of blood, urine and CSF biomarkers of PD pathology
  Interventions: Other: Positron Emission Tomography (PET) scan using BU99008 tracer; Other: FP-CIT Single-photon Emission Computed Tomography (SPECT) scan; Other: Magnetic Resonance Imaging (MRI) Scan; Other: Lumbar puncture
- Healthy Control: PET and SPECT molecular imaging and MRI; Clinical investigation and computerized neuropsychological testing; Collection of blood, urine and CSF biomarkers of PD patholog
  Interventions: Other: Positron Emission Tomography (PET) scan using BU99008 tracer; Other: FP-CIT Single-photon Emission Computed Tomography (SPECT) scan; Other: Magnetic Resonance Imaging (MRI) Scan; Other: Lumbar puncture

INTERVENTIONS:
Other: Positron Emission Tomography (PET) scan using BU99008 tracer — A positron emission tomography (PET) scan produce detailed 3-dimensional images of the inside of the body by showing radiation from tracers used to highlight specific areas of the brain.
Other: FP-CIT Single-photon Emission Computed Tomography (SPECT) scan — A single-photon emission computerized tomography (SPECT) scan allows analysis of brain function by creating 3D Pictures using compounds called tracers.
Other: Magnetic Resonance Imaging (MRI) Scan — MRI (magnetic resonance imaging) uses magnets alongside radio waves to create pictures of the brain.
Other: Lumbar puncture — A lumbar puncture is where a thin needle is inserted between the bones in your lower spine using local anaesthetic. This allows the collection of Cerebrospinal fluid ( CSF)

SUMMARY:
In this study, the researchers aim to find a biomarker of PD. Using imaging scans called Positron Emission tomography (PET), Single Photon Emission Computed Tomography (SPECT), and Magnetic Resonance Imaging (MRI). The PET and SPECT scans use small amounts of radiation and specific compounds called tracers, to study chemical changes in the brain in a way not possible with any other procedure. The MRI uses magnetic fields to generate images of brain structure and function

DETAILED DESCRIPTION:
Parkinson's disease is a chronic neurological disease that progresses over time and causes a variety of symptoms, such as slowness of movement, stiffness and shaking. The purpose of this study is to find a biomarker for Parkinson's disease. A biomarker is an indicator of the presence of a disease, that can be measured, and that is able to give information.

The study will take place in London, in three research sites that are located near to each other. The NIHR Imperial Clinical Research Facility (CRF) at Hammersmith Hospital in London, for clinical assessment, and Invicro London for imaging assessments. Both Hammersmith Hospital and Invicro are located at Hammersmith Hospital Campus.

Taking part in this study will involve two sets of visits spaced out 12 months apart. These visits would include, initial screening and consent visit. The second visit would be for an MRI and PET scan with the tracer BU99008 which highlights astroglia cells. The third visit would be for a SPECT scan, and an optional fourth visit for a Lumbar Puncture procedure to collect spinal fluid for analysis.

These visits are then repeated 12 months later to form a comparison. The maximum number of visits for this study would be 8, however two of these visits are optional lumbar puncture visits.

The findings form this research will provide a deeper understanding of the brain changes in Parkinson's disease. More importantly, this study will help with the discovery and development of new medications aiming to delay progression of Parkinson's disease symptoms. n about the progression, or severity, of it.

ELIGIBILITY:
Inclusion criteria

* All subjects must be judged by the investigator able to understand the nature, design, and procedures of the study and must be able to provide a signed and dated informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations.
* All subjects must be willing and able to comply with scheduled visits, required study procedures and laboratory tests.
* All subjects must be able to travel to the research sites for the study procedures.
* Age 25 years or older.
* For female subjects: They must be either of non-childbearing potential (either surgically sterile or post- menopausal - defined as 12 months of spontaneous amenorrhea), or, if of childbearing potential, subjects must demonstrate to be non-pregnant (as demonstrated by negative urine β-HCG test at screening), non-breastfeeding.
* All subjects must comply with highly effective contraceptive measures. A highly effective contraceptive measure is defined as a measure that can achieve a failure rate of less than 1% per year when used consistently and correctly. These methods are listed in more detail below:

Oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation;

Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation:

Intrauterine device (IUD)

Intrauterine hormone-releasing system (IUS)

Bilateral tubal occlusion

Vasectomised partner

Sexual abstinence

* For sexually active male subjects, they must agree to use condoms to protect their partners from becoming pregnant for the duration of the study and for 3 months after the last administration of PET or SPECT ligands. They must also agree to ensure that they and their partners are routinely using a medically approved contraceptive method. It is important that male subjects not impregnate others for the duration of the study and for 3 months after the last administration of PET or SPECT ligands.
* All subjects must have adequate visual and auditory acuity according to investigator's judgement to complete the psychological testing.
* All subjects must have no use of medications with known interaction with I2BS (e.g. idaxozan, efaroxan, yohimbine, atomoxetine, atipamezole, mianserin, mirtazapine, clonidine, guanfacine, guanabenz, guanethidine, xylazine, tizanidine, tedetomidine, methyldopa, fadolmidine, dexmedetomidine)
* For subjects taking any drugs that might interfere with dopamine transporter SPECT imaging (neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative) must be willing and able from a medical standpoint to hold the medication for at least 5 half-lives prior to screening DaTSCANä imaging.

Exclusion criteria

* Subjects lacking capacity according to investigator's judgment;
* Subjects with a clinical diagnosis of dementia as determined by the investigator;
* Subjects with current or a recent history of drug or alcohol abuse/dependence;
* Current treatment with anticoagulants (e.g. warfarin, heparin) that might preclude the arterial cannulation and the safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Negative Allen test in both hands,
* Use of any of the following drugs that might interfere with dopamine transporter SPECT imaging: neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative, within 5 months of Screening.
* Use of any medications with known actions on I2BS (e.g. idaxozan, efaroxan, yohimbine, atomoxetine, atipamezole, mianserin, mirtazapine, clonidine, guanfacine, guanabenz, guanethidine, xylazine, tizanidine, tedetomidine, methyldopa, fadolmidine, dexmedetomidine);
* Use of investigational drugs or devices within 60 days prior to Baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).
* History of cancer within the last 5 years, with the exception of non-metastatic basal cell carcinoma of the skin.
* Subjects with current or recent history of drug or alcohol abuse/dependence.
* Contraindication to MRI, such as presence of metal devises or implants (e.g. pacemaker, vascular- or heart- valves, stents, clips), metal deposited in the body (e.g. bullets or shells), or metal grains in the eyes;
* Claustrophobia or history of back pain that makes prolonged laying on the PET, SPECT, or MRI scanner intolerable.
* Previously obtained MRI scan with evidence of clinically significant neurological disorder (in the opinion of the Investigator).
* Presence of any clinically significant medical condition (including cardiovascular, respiratory, cerebrovascular, hematological, hepatic, renal, gastrointestinal, or other disease) that, based on the judgment of the investigator, is clinically unstable, is likely to deteriorate during the course of the study, could put the patient at risk because of participation in the study, could affect the subject's ability to complete the study, or could influence the study results;
* History of suicidal behavior or active suicidal ideation;
* Pregnancy or breastfeeding or intent to become pregnant in the next 18 months;

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of carriers of SNCA genetic mutations for familial forms of Parkinson's Disease, idiopathic Parkinson's Disease patients and previously collected data from healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PET scan with BU99008 to highlight I2BS and and Astroglia cells. | 12 Months
  This used to show the role of Astroglia cell activation in Parkinson's disease to understand the role of Astroglia in Parkinson's disease Pathophysiology
Single Photon Emission Computed Tomography (SPECT) to measure brain molecular pathology | 12 Months
  To quantify serotonergic pathology with BU99008 and dopaminergic pathology with Single-photon Emission Computed Tomography (SPECT)
Magnetic Resonance Imaging (MRI) | 12 Months
  Magnetic Resonance Imaging (MRI) to view structural and microstructural changes and structural connectivity..

OTHER OUTCOMES:
Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 12 Months
  To determine if there is a correlation with neuropsychological and behavioural evaluation.
Montreal Cognitive Assessment (MOCA) to determine if there is a correlation with neuropsychological and behavioural evaluation | 12 Months
  A cognitive screening test designed to assist in the detection of mild cognitive impairment, scored out of 30
Cambridge Neuropsychological Test Automated Battery (CANTAB) to determine if there is a correlation with neuropsychological and behavioural evaluation | 12 Months
  Administered to detect cognitive issues & brain disorders efficiently.
Symbol Digit Modalities Test (SDMT) to determine if there is a correlation with neuropsychological and behavioural evaluation | 12 Months
  To be used in screening for organic cerebral dysfunction scored out of 110
Beck Depression Inventory-II (BDI-II) to determine if there is a correlation with neuropsychological and behavioural evaluation | 12 Months
  A brief, self-report inventory designed to measure the severity of depression symptomatology
State-Trait Anxiety Inventory (STAI) to determine if there is a correlation with neuropsychological and behavioural evaluation | 12 Months
  A commonly used measure of trait and state anxiety. Used to diagnose anxiety and to distinguish it from depressive syndromes
University of Pennsylvania Smell Identification Test (UPSIT) to determine if there is a correlation with neuropsychological and behavioural evaluation | 12 Months
  This is used to test the function of an individual's olfactory system
Movement Disorder Society- Non-Motor Symptoms scale for Parkinson's Disease MDS-NMSS to determine if there is a correlation with neuropsychological and behavioural evaluation | 12 Months
  This is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease
Scales for Outcomes in Parkinson's Disease-Autonomic questionnaire - Autonomic Dysfunction (SCOPA-AUT) to determine if there is a correlation with neuropsychological and behavioural evaluation | 12 Months
  A 25 item assessment to evaluate autonomic symptoms in patients with Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Marios Politis, Professor, Principal Investigator — University of Exeter
Locations (1):
- University Of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Yet to be confirmed

REFERENCES:
- See also: University of Exeter brief project information webpage — https://medicine.exeter.ac.uk/clinical-biomedical/research/nig/currentstudies/